CLINICAL TRIAL: NCT00056784
Title: The Pathogenesis of Chronic Graft Failure After Kidney Transplantation
Brief Title: The Role of Connective Tissue Growth Factor in the Development of Kidney Disease After Organ Transplantation
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030132; 03-DK-0132
Record Dates: First submitted 2003-03-22; First posted 2003-03-24 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2014-06-17

CONDITIONS: Kidney Transplantation
Keywords: TGF-Beta; Kidney; Transplantation; Rejection; Immunosuppression; Kidney Transplant; Chronic Allograft Nephropathy; CAN
MeSH Terms: conditions — Camurati-Engelmann Syndrome; Rejection, Psychology

SUMMARY:
This study will examine whether measurements of connective tissue growth factor (CTGF) and other cell proteins can identify which kidney transplant recipients are likely to develop chronic allograft nephropathy (CAN), a disease of the transplanted kidney. CAN may occur months to years after the transplant. The kidney becomes progressively scarred and eventually loses all function, so that dialysis or another transplant is needed. A better understanding of how CTGF and other proteins are involved in the development of CAN may provide new targets for treating for the disease.

Patients who are scheduled to receive a kidney or combined kidney-pancreas transplant or who have received a transplant recently (within 6 months) may be eligible for this study. Participants will be enrolled before the transplant, if possible, or after the transplant, and will undergo the following tests and procedures:

* Physical examinations at the screening visit, at 1, 6, 12, and 24 months, and then once yearly.
* Blood sample collections at the screening visit, at 1, 6, 12, 18, and 24 months and then once yearly.
* Urine sample collections at the screening visit, at 1, 6, 12, 18, and 24 months and then once yearly.
* Kidney biopsies at the beginning of the study, at 1, 6, 12, and 24 months, and then once a year for research purposes. Participants may refuse to have a research biopsy at any time during the study. Also, patients who are having a kidney biopsy for another reason at these time points will not have a second biopsy. The biopsy procedure takes about 15 minutes and is done in the hospital. The patient lies on his or her back and the skin over the transplanted kidney is cleaned with alcohol and iodine. The area is numbed with an injection of an anesthetic, and then a biopsy needle is placed through the kin. The biopsy may be repeated up to three times to get enough tissue to test for CAN. Patients lie flat for 4 hours after the procedure to reduce the risk of bleeding, and are observed for another 2 hours for possible complications.

DETAILED DESCRIPTION:
Following transplantation, recipients of organ allografts are placed on immunosuppression indefinitely. Despite dramatic improvements in acute rejection rates and short-term graft survival, long term graft survival has not changed appreciably over the past 20 years. In kidney transplantation, the leading cause of late graft loss is chronic allograft nephropathy (CAN). This disorder is clinically characterized by a progressive decline in kidney function, associated with the characteristic histologic features of interstitial fibrosis and inflammation, arteriosclerosis, glomerulosclerosis, and tubular atrophy. Both immunologic and non-immunologic factors have been implicated in the development of CAN. However, the etiology of this disorder has not been clearly defined nor is there specific therapy for treating CAN.

Implicated in the development of CAN in rodents and humans is transforming growth factor beta (TGF-beta), a pleiotropic cytokine which is elevated in CAN recipients, and stimulates matrix deposition within the graft. A downstream effector of TGF-b is connective tissue growth factor (CTGF), which has been recently associated with other fibrotic renal diseases. In preliminary studies in a mouse model of CAN, CTGF gene expression is increased in kidney transplants with CAN. However, its role in human CAN is unknown.

The aim of this investigation is to identify whether CTGF may play a role in the pathogenesis of CAN in humans. Our long-term objective is to determine whether CTGF and other cytokine mediators may be novel targets for the therapy of CAN. Our goals are to: 1. Determine the level of CTGF expressed in the urine and serum CTGF of recipients of kidney transplants; 2. Identify whether urinary or serum CTGF might be a marker of CAN and be utilized as a predictor for those at risk to develop the disease; 3. Identify other molecular messages and proteins that may identify the development of CAN, as potential future targets of treatment.

In this prospective study, serial urine and serum samples will be obtained in recipients, before, during, and after transplantation of a kidney allograft. The graft will be monitored in the context of standard measures of renal function, which include serum creatinine and creatinine clearance. These results will be correlated with other clinically descriptive information regarding the recipient s transplant.

ELIGIBILITY:
* INCLUSION CRITERIA:

Recipients of living related, living unrelated, and cadaveric kidney transplants.

This study will be open to all patients currently enrolled in NIDDK transplant protocols as well as patients recruited from other transplant centers.

Ability and willingness to provide informed consent (adults greater than or equal to 18.0 years) or assent (children 4 to 18.0 years).

EXCLUSION CRITERIA:

Inability to provide informed consent.

Inability to return to NIH for follow-up.

Inability or unwillingness to release outside medical records or pathology.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2003-03-20; Study Completion 2014-06-17

CONTACTS AND LOCATIONS:
Overall Officials: Monique E Cho, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wolfe RA, Ashby VB, Milford EL, Ojo AO, Ettenger RE, Agodoa LY, Held PJ, Port FK. Comparison of mortality in all patients on dialysis, patients on dialysis awaiting transplantation, and recipients of a first cadaveric transplant. N Engl J Med. 1999 Dec 2;341(23):1725-30. doi: 10.1056/NEJM199912023412303. PMID 10580071
- [Background] Hariharan S, Johnson CP, Bresnahan BA, Taranto SE, McIntosh MJ, Stablein D. Improved graft survival after renal transplantation in the United States, 1988 to 1996. N Engl J Med. 2000 Mar 2;342(9):605-12. doi: 10.1056/NEJM200003023420901. PMID 10699159
- [Background] Cecka JM. The UNOS renal transplant registry. Clin Transpl. 2001:1-18. PMID 12211771